CLINICAL TRIAL: NCT02825498
Title: Randomised Prospective Trial Comparing Contact Force and Non-contact Force Guided Catheter Ablation for Cavotricuspid Isthmus Dependent Atrial Flutter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Victoria Cardiac Arrhythmia Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C2016-012
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Atrial Flutter; Radiofrequency Catheter Ablation
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Operator guided by contact force (Experimental): Operator has full access to contact force parameters including force time integral (FTI).
  Interventions: Device: Contact force guided RFA
- Operator blinded to contact force (No Intervention): Operator is blinded to contact force with ablation guided by standard markers of effective ablation.

INTERVENTIONS:
Device: Contact force guided RFA — Contact force guided RFA during Atrial Flutter ablation procedure.
  Arms: Operator guided by contact force

SUMMARY:
Radiofrequency ablation (RFA) is a standard treatment option for cavotricuspid isthmus (CTI) dependent atrial flutter. We plan to perform a randomized prospective trial comparing the efficacy of contact force (CF) guided CTI ablation against catheter ablation with the operator blinded to contact force parameters.

DETAILED DESCRIPTION:
Subjects will be followed for one year post procedure in order to check for atrial flutter recurrences. This will involve an in-person visit at 3 months post procedure, and records checks at 12 months post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over the age of 18) with 12 lead ECG documented paroxysmal or persistent CTI dependent atrial flutter planned to undergo CTI ablation.
* Able and willing to give informed consent.

Exclusion Criteria:

* Previous CTI ablation
* Previous non-CTI dependent atrial flutter (ie.patients with previous history of pulmonary vein isolation or left atrial ablation, congenital heart disease, surgical ablation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-05-18 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of RFA | Determined during RFA procedure
  Total RFA time required to achieve bidirectional block

SECONDARY OUTCOMES:
Recurrence of atrial flutter | Assessed at 12 weeks and 12 months post CTI RFA procedure
  Documented recurrence of atrial flutter
Average total CF achieved | Determined during RFA procedure
  Average total CF per ablation per segment (third) of the CTI.
Average axial CF achieved | Determined during RFA procedure
  Average axial CF per ablation per segment (third) of the CTI.
Average FTI achieved | Determined during RFA procedure
  Average FTI per ablation per segment (third) of the CTI.
Average lateral CF achieved | Determined during RFA procedure
  Average lateral CF per ablation per segment (third) of the CTI.
Average lesion size index (LSI) achieved | Determined during RFA procedure
  Average lesion size index (LSI) per ablation per segment (third) of the CTI.
Procedural complication rate | Determined during RFA procedure and at 12 weeks post RFA procedure
  Incidence of procedural complications: stroke, cardiac perforation, steam pops, access site bleeding.
Average total CF of segment of acute and delayed reconnection | Determined during index and repeat RFA procedure
  Average total CF per ablation in segment (third) of acute or delayed reconnection.
Average lateral CF of segment of acute and delayed reconnection | Determined during index and repeat RFA procedure
  Average lateral CF per ablation in segment (third) of acute or delayed reconnection.
Average axial CF of segment of acute and delayed reconnection | Determined during index and repeat RFA procedure
  Average axial CF per ablation in segment (third) of acute or delayed reconnection.
Average FTI of segment of acute and delayed reconnection | Determined during index and repeat RFA procedure
  Average FTI per ablation in segment (third) of acute or delayed reconnection.
Average lesion size index (LSI) of segment of acute and delayed reconnection | Determined during index and repeat RFA procedure
  Average lesion size index (LSI) per ablation in segment (third) of acute or delayed reconnection.
Procedural efficacy of RFA | Determined during RFA procedure
  Total procedural time required to achieve bidirectional block

CONTACTS AND LOCATIONS:
Overall Officials: Paul Novak, MD, Principal Investigator — Victoria Cardiac Arrhythmia Trials
Locations (1):
- Victoria Cardiac Arrhythmia Trials, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
De-identified IPD may be shared with other researchers upon study completion. Data may be obtained by contacting Victoria Cardiac Arrhythmia Trials Inc. at 250-595-0400.